CLINICAL TRIAL: NCT05709964
Title: Comparison of Demographic Data Mentioned by the Patients or Measured by a Physician
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, FAACD, Head of Department, Astes
Other Study IDs: PTS
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Self Report

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All patients included in this study. Investigators will record both self-reported and measured height, weight, and neck circumference in all of these patients.
  Interventions: Other: Self-reported; Other: Measured

INTERVENTIONS:
Other: Self-reported — Self-reported height, weight, and neck circumference
Other: Measured — Height, weight, and neck circumference measured by the investigator.

SUMMARY:
OSA (Obstructive Sleep Apnea) represents a major risk of postoperative complications. Predictive scores have been developed as the STOP-Bang score and the DES-OSA score. These scores take into account morphological parameters such as weight, height, and neck circumference. These data can be contained from the patients (self-reported) or by the measurements performed by a physician. The aim of this study is to compare the accuracy of both measurements (self-reported by the patient or measured by the physicians).

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective surgery on a one-day hospital

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients included
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of self-reported height measurements | One month
  The aim of this study is to determine the accuracy of the self-reported height (compared to height measured by the physician).
Accuracy of self-reported weight measurements | One month
  The aim of this study is to determine the accuracy of the self-reported weight (compared to height measured by the physician).
Accuracy of self-reported neck circumference measurements | One month
  The aim of this study is to determine the accuracy of the self-reported neck circumference (compared to height measured by the physician).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, PhD, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No